CLINICAL TRIAL: NCT05174208
Title: Study of Imaginomics Predicting Early Surgical Rates in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-ZSLYEC-341
Record Dates: First submitted 2021-09-24; First posted 2021-12-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease; Prognostic Model; Radiomics
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD
  Interventions: Other: CTE examination

INTERVENTIONS:
Other: CTE examination — each patients should have undergone CTE examination

SUMMARY:
Crohn's disease (CD), a type of inflammatory bowel disease (IBD), is a chronic intestinal recurrent inflammatory disease involving the entire digestive tract. Most CD patients require surgery for complications, including stenosis, perforation, and severe intestinal bleeding. Predicting early-onset surgery risk is of great importance to assist launching of therapeutic strategies. We aim to establish a digital prognostic model and nomogram using radiomics, which will help clinical practice.

ELIGIBILITY:
Inclusion Criteria:

patients with a confirmed diagnosis of CD; a follow-up more than 1 year; without previous CD-associated intestinal surgeries; complete data of CTE.

Exclusion Criteria:

patients without a confirmed diagnosis of CD; with incomplete data and a follow-up less than 1 year; patients have previous intestinal surgeries; patients who have never undergone CTE examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2017-2020 CD patients in the IBD center of Sixth Affiliated Hospital of Sun Yat-Sen University.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
percentages of surgery at one-year after diagnosis | 2017-2021
  percentages of surgery at one-year after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China